CLINICAL TRIAL: NCT05816954
Title: Artificial Intelligence-based Identification of Imaging Biomarkers of Lung FRAILty in Patients With Acute Respiratory Distress Syndrome.
Brief Title: Imaging Biomarkers to Stratify the Risk of Barotrauma in ARDS
Acronym: FRAIL ARDS
Status: Recruiting | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Full Professor, Università Vita-Salute San Raffaele
Other Study IDs: FRAIL ARDS - 49/INT/2022
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome; Barotrauma
MeSH Terms: conditions — Respiratory Distress Syndrome; Barotrauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Chest Computed Tomography Scan per normal clinical practice — Normal Clinical practice

SUMMARY:
The high incidence of barotrauma in patients with COVID-19-related acute respiratory distress syndrome (ARDS) (16.1%, with a mortality rate >60%) provides rationale for considering COVID-19 ARDS a paradigm for lung frailty. The investigators recently discovered that the Macklin effect is an impressive radiological predictor of barotrauma in COVID-19 ARDS. Since lung frailty is a major issue also in non-COVID-19 ARDS (6% barotrauma, with a mortality rate of 46% ) the investigators want to confirm the importance of Macklin effect in non-COVID-19 ARDS. Using artificial intelligence-based approaches the investigators also want to identify imaging biomarkers to non-invasively assess lung frailty in a mixed cohort of COVID-19/non-COVID-19 ARDS patients. Furthermore, the investigators want to prospectively validate these biomarkers in a cohort of ARDS patients. This will provide a therapeutic algorithm for ARDS patients at high-risk for barotrauma, identifying those most likely to benefit from hyper protective strategies.

DETAILED DESCRIPTION:
Development of barotrauma, spanning from asymptomatic air leakage within lung parenchyma to life-threatening conditions such as tension pneumothorax, is frequent in acute respiratory distress syndrome (ARDS), with a difficult, non-standardized management, resulting in high mortality rates (greater than 60% in coronavirus disease 2019 [COVID-19] ARDS patients, around 46% in non-COVID-19 ARDS patients). Of note, barotrauma occurs also in spontaneously breathing patients with COVID-19 ARDS. Frailty of lung parenchyma represents indeed a major issue in ARDS. In addition, in high-risk patients, mechanical ventilation may exacerbate pulmonary damage (ventilator-induced lung injury) and potentially induce barotrauma despite use of protective mechanical ventilation. Early assessment of lung frailty could therefore allows early risk stratification in terms of barotrauma susceptibility amongst ARDS patients, providing rationale for the deployment of lung protective management strategies in those at high-risk for barotrauma. Macklin effect, firstly intended to allow proper differentiation between respiratory and other causes of air leakage in the mediastinum (such as tracheobronchial/oesophageal injury), has been recently proved by our group to be a consistent, very accurate radiological predictor of barotrauma development in COVID-19 ARDS patients (sensitivity: 89.2%; specificity: 95.6%), anticipating by 12 days the occurrence of clinically overt barotrauma. These results have been confirmed, and even improved by multicentre findings, which report, on a large cohort of COVID-19 patients (almost 700), an impressive, almost perfect overall accuracy (99.8%) of the Macklin effect in predicting barotrauma development. Furthermore, data from our group suggest that early application of awake veno/venous extracorporeal membrane oxygenation (ECMO) without invasive mechanical ventilation in COVID-19 severe ARDS patients at high-risk for barotrauma (those with Macklin effect on chest CT imaging) is feasible and may result in no barotrauma events and low intubation rate. In this respect, confirmation of Macklin effect role and identification of further, novel quantitative imaging biomarkers could unveil biological bases of lung frailty in course of ARDS and provide instruments for early risk stratification before barotrauma occurrence.

Our group also implemented original in-house facilities consisting of densitometry, machine learning and artificial intelligence-based approaches to assess lung composition in COVID-19 patients throughout a fully automated workflow; recently, the investigators highlighted the outstanding clinical significance of this methodological approach in predicting patients' prognosis, as well as its great reproducibility. Preliminary, yet unpublished findings suggest that lung frailty has a specific densitometric signature, being a possible marker for hyper protective management strategies; few, highly robust radiomic features seem to corroborate the same result.

Accordingly, the driving hypotheses of this retrospective/prospective study are that, irrespective of COVID-19 status, in ARDS patients, i) lung frailty has a specific pattern of imaging biomarkers, and that ii) a more accurate selection of patients could limit the problem of barotrauma associated with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological signs of ARDS, according to Berlin criteria [14], requiring ICU admission;
* Obtain duly signed informed consent.

Exclusion Criteria:

* Poor quality imaging (because of motion/respiratory artefacts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS clinical suspicion or diagnosis will be enrolled; specifically, these patients will be admitted at intensive care unit. All patients enrolled in the prospective cohort will follow their normal course of diagnosis/treatment without any further requirements for the scope of this study other than those provided in the normal management of patients with this condition. Furthermore, any decision regarding drug or procedure will be made by the physician based on her/his clinical judgment in the context of clinical practice, independently from the decision to include the patient in this study. No follow-up medical and/or imaging examinations/laboratory analysis after hospital discharge are needed by the present study design.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically relevant barotrauma | 30 days or until hospital discharge. Specifically, from date of basal CT scan until the date of first radiologically documented barotrauma.
  Barotrauma is diagnosed only in the case of clear radiological evidence (free air at chest X-ray and/or chest CT scan).
  When a "central" (non-alveolar) cause of barotrauma (tracheal fissure, esophageal rupture) is suspected, endoscopy will be performed.
  Patients with barotrauma occurring within twelve hours from a chest interventional procedure (e.g. drains placement, central venous catheters insertion) will be excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, Professor, Study Chair — Vita-Salute San Raffaele University
Locations (2):
- Italy (2):
  - Ospedale Mater Domini, Catanzaro, Calabria
  - IRCCS San Raffaele Scientific Institute, Milan, MI

REFERENCES:
- [Background] Belletti A, Todaro G, Valsecchi G, Losiggio R, Palumbo D, Landoni G, Zangrillo A. Barotrauma in Coronavirus Disease 2019 Patients Undergoing Invasive Mechanical Ventilation: A Systematic Literature Review. Crit Care Med. 2022 Mar 1;50(3):491-500. doi: 10.1097/CCM.0000000000005283. PMID 34637421
- [Background] Palumbo D, Campochiaro C, Belletti A, Marinosci A, Dagna L, Zangrillo A, De Cobelli F; COVID-BioB Study Group. Pneumothorax/pneumomediastinum in non-intubated COVID-19 patients: Differences between first and second Italian pandemic wave. Eur J Intern Med. 2021 Jun;88:144-146. doi: 10.1016/j.ejim.2021.03.018. Epub 2021 Mar 19. No abstract available. PMID 33820685
- [Background] Sakai M, Murayama S, Gibo M, Akamine T, Nagata O. Frequent cause of the Macklin effect in spontaneous pneumomediastinum: demonstration by multidetector-row computed tomography. J Comput Assist Tomogr. 2006 Jan-Feb;30(1):92-4. doi: 10.1097/01.rct.0000187416.07698.8d. PMID 16365580
- [Background] Murayama S, Gibo S. Spontaneous pneumomediastinum and Macklin effect: Overview and appearance on computed tomography. World J Radiol. 2014 Nov 28;6(11):850-4. doi: 10.4329/wjr.v6.i11.850. PMID 25431639
- [Background] Russell DW, Watts JR Jr, Powers TA. Searching for the Source of the Leak: PIE and the Macklin Effect. Ann Am Thorac Soc. 2018 Nov;15(11):1354-1356. doi: 10.1513/AnnalsATS.201803-200CC. No abstract available. PMID 30382777
- [Background] Belletti A, Palumbo D, Zangrillo A, Fominskiy EV, Franchini S, Dell'Acqua A, Marinosci A, Monti G, Vitali G, Colombo S, Guazzarotti G, Lembo R, Maimeri N, Faustini C, Pennella R, Mushtaq J, Landoni G, Scandroglio AM, Dagna L, De Cobelli F; COVID-BioB Study Group. Predictors of Pneumothorax/Pneumomediastinum in Mechanically Ventilated COVID-19 Patients. J Cardiothorac Vasc Anesth. 2021 Dec;35(12):3642-3651. doi: 10.1053/j.jvca.2021.02.008. Epub 2021 Feb 6. PMID 33678544
- [Background] Palumbo D, Zangrillo A, Belletti A, Guazzarotti G, Calvi MR, Guzzo F, Pennella R, Monti G, Gritti C, Marmiere M, Rocchi M, Colombo S, Valsecchi D, Scandroglio AM, Dagna L, Rovere-Querini P, Tresoldi M, Landoni G, De Cobelli F; COVID-BioB Study Group. A radiological predictor for pneumomediastinum/pneumothorax in COVID-19 ARDS patients. J Crit Care. 2021 Dec;66:14-19. doi: 10.1016/j.jcrc.2021.07.022. Epub 2021 Aug 12. PMID 34392131
- [Background] Paternoster G, Belmonte G, Scarano E, Rotondo P, Palumbo D, Belletti A, Corradi F, Bertini P, Landoni G, Guarracino F; COVID-Macklin Study Group. Macklin effect on baseline chest CT scan accurately predicts barotrauma in COVID-19 patients. Respir Med. 2022 Jun;197:106853. doi: 10.1016/j.rmed.2022.106853. Epub 2022 Apr 20. PMID 35512457
- [Background] Paternoster G, Bertini P, Belletti A, Landoni G, Gallotta S, Palumbo D, Isirdi A, Guarracino F. Venovenous Extracorporeal Membrane Oxygenation in Awake Non-Intubated Patients With COVID-19 ARDS at High Risk for Barotrauma. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt B):2975-2982. doi: 10.1053/j.jvca.2022.03.011. Epub 2022 Mar 17. PMID 35537972
- [Background] Mori M, Palumbo D, De Lorenzo R, Broggi S, Compagnone N, Guazzarotti G, Giorgio Esposito P, Mazzilli A, Steidler S, Pietro Vitali G, Del Vecchio A, Rovere Querini P, De Cobelli F, Fiorino C. Robust prediction of mortality of COVID-19 patients based on quantitative, operator-independent, lung CT densitometry. Phys Med. 2021 May;85:63-71. doi: 10.1016/j.ejmp.2021.04.022. Epub 2021 Apr 30. PMID 33971530
- [Background] Mori M, Alborghetti L, Palumbo D, Broggi S, Raspanti D, Rovere Querini P, Del Vecchio A, De Cobelli F, Fiorino C. Atlas-based lung segmentation combined with automatic densitometry characterization in COVID-19 patients: Training, validation and first application in a longitudinal study. Phys Med. 2022 Aug;100:142-152. doi: 10.1016/j.ejmp.2022.06.018. Epub 2022 Jul 4. PMID 35839667
- [Background] Palumbo D, Mori M, Prato F, Crippa S, Belfiori G, Reni M, Mushtaq J, Aleotti F, Guazzarotti G, Cao R, Steidler S, Tamburrino D, Spezi E, Del Vecchio A, Cascinu S, Falconi M, Fiorino C, De Cobelli F. Prediction of Early Distant Recurrence in Upfront Resectable Pancreatic Adenocarcinoma: A Multidisciplinary, Machine Learning-Based Approach. Cancers (Basel). 2021 Sep 30;13(19):4938. doi: 10.3390/cancers13194938. PMID 34638421
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452